CLINICAL TRIAL: NCT02269605
Title: Bryostatin-1 Effect on HIV-1 Latency and Reservoir HIV-1 Infected Patients Receiving Antiretroviral Treatment: Pilot, Controlled, Double Blinded, Dose Searching Trial
Brief Title: Bryostatin-1 Effect on HIV-1 Latency and Reservoir in HIV-1 Infected Patients Receiving Antiretroviral Treatment
Acronym: BRYOLAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRYOLAT
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infection
Keywords: HIV reservoir; Bryostatin
MeSH Terms: conditions — HIV Infections | interventions — bryostatin 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Placebo Comparator): Patients receiving placebo (sodium chloride) at single dose
  Interventions: Other: Placebo
- Group 2 (Active Comparator): Patients receiving Bryostatin 1 (10ug/m2) at single dose
  Interventions: Drug: Bryostatin 1 (10ug/m2)
- Group 3 (Active Comparator): Patients receiving Bryostatin 1 (20ug/m2) at single dose
  Interventions: Drug: Bryostatin 1 (20ug/m2)

INTERVENTIONS:
Other: Placebo — Group 1: Placebo (sodium chloride 0.8 %) at single dose
  Arms: Group 1
Drug: Bryostatin 1 (10ug/m2) — Group 2: Bryostatin 1 (10ug/m2) at single dose
  Arms: Group 2
Drug: Bryostatin 1 (20ug/m2) — Group 3: Bryostatin 1 (20ug/m2) at single dose
  Arms: Group 3

SUMMARY:
Phase I, randomized, double blind, placebo-controlled, dose-finding trial. The trial´s goal is to evaluate two different doses of Bryostatin on HIV-1 latency and reservoir in HIV-1 infected patients receiving antiretroviral treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients understanding the trial purpose
* Patients between 18 and 50 years of age
* Patients with chronic HIV-1 infection
* Patients receiving antiretroviral treatment with at least 3 active drugs for at least 2 years
* Undetectable viral load measured by ultra sensitive methods
* CD4+ levels higher than 350 cells/mm3
* Patients committed to use contraceptive methods during the trial and up to 3 months after.

Exclusion Criteria:

* Previous antiretroviral treatment failure, as any viral load outbreak after having had undetectable HIV-1 load. Low grade, transitory outbreaks (<200 RNA copies/ml) resolved without treatment modifications are excluded
* Patients planned to interrupt antiretroviral treatment during the trial
* Patients receiving immunosuppressant or immunostimulant drugs, including valproic acid.
* Pregnant women
* Bryostatin-1 hypersensitivity
* Being enrolled in another clinical trial or having participated in another clinical trial in the previous 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intracellular HIV-1 RNA (usRNA and msRNA) level before and after bryostatin-1 administration | Baseline visit and days 2 and 3 after the day of treatment

SECONDARY OUTCOMES:
HIV-1 RNA level | Baseline visit, day 0 (15, 30, 60 minutes after begining of drug administration and 1, 2, 4, 8, 12 hours after begining of drug administration) and days 1, 2 and 3
CD4+ and CD8+ T (CD38+ and HLA DR+ positive) cell level | Baseline visit, day 1 and day 3
Episomal DNA with 2 LTRs level | Baseline visit, day 1 and day 3
Adverse Events | From baseline visit to day 28 after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Moreno, MD, PhD, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Infectious Diseases Service, Madrid, Non US/Canada, Spain

REFERENCES:
- [Background] Persaud D, Zhou Y, Siliciano JM, Siliciano RF. Latency in human immunodeficiency virus type 1 infection: no easy answers. J Virol. 2003 Feb;77(3):1659-65. doi: 10.1128/jvi.77.3.1659-1665.2003. No abstract available. PMID 12525599
- [Background] Blankson JN, Gallant JE, Quinn TC, Bartlett JG, Siliciano RF. Loss of HIV-1-specific immunity during treatment interruption in 2 chronically infected patients. JAMA. 2002 Jul 10;288(2):162-4. doi: 10.1001/jama.288.2.162-a. No abstract available. PMID 12095377
- [Background] Richman DD, Margolis DM, Delaney M, Greene WC, Hazuda D, Pomerantz RJ. The challenge of finding a cure for HIV infection. Science. 2009 Mar 6;323(5919):1304-7. doi: 10.1126/science.1165706. PMID 19265012
- [Derived] Gutierrez C, Serrano-Villar S, Madrid-Elena N, Perez-Elias MJ, Martin ME, Barbas C, Ruiperez J, Munoz E, Munoz-Fernandez MA, Castor T, Moreno S. Bryostatin-1 for latent virus reactivation in HIV-infected patients on antiretroviral therapy. AIDS. 2016 Jun 1;30(9):1385-92. doi: 10.1097/QAD.0000000000001064. PMID 26891037